CLINICAL TRIAL: NCT00457002
Title: A Phase 3 Randomized, Double-Blind, Parallel-group, Multi-center Study of the Safety and Efficacy of Apixaban for Prophylaxis of Venous Thromboembolism in Acutely Ill Medical Subjects During and Following Hospitalization.
Brief Title: Study of Apixaban for the Prevention of Thrombosis-related Events in Patients With Acute Medical Illness
Acronym: ADOPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-036
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2014-05

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Prevention of deep vein thrombosis and pulmonary embolism with acutely ill hospitalized patients
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — apixaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): While hospitalized, Apixaban plus Placebo
  Apixaban (Tablets, Oral, 2.5 mg), Placebo (Syringes, SC)
  After hospital discharge, Apixaban
  Apixaban (Tablets, Oral, 2.5 mg)
  Interventions: Drug: Apixaban
- Arm 2 (Active Comparator): While hospitalized, Enoxaparin plus Placebo
  Enoxaparin (Syringes, SC, 40 mg), Placebo (Tablets, Oral)
  After hospital discharge: Placebo
  Placebo (Tablets, Oral)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Apixaban — Apixaban: Twice daily, 30 days
  Placebo: Once daily, 6-14 days
  Other Names: BMS-562247
  Arms: Arm 1
Drug: Enoxaparin — Enoxaparin: Once daily, 6-14 days
  Placebo: Twice daily, 30 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to learn if apixaban can prevent blood clots in the leg (deep vein thrombosis [DVT]) and lung (pulmonary embolism [PE]) that sometimes occur within patients hospitalized for acute medical illness, and to learn how apixaban compares to enoxaparin (Lovenox®) for preventing these clots. The safety of apixaban will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant, non-breastfeeding women
* 40 years or older
* hospitalized with congestive heart failure or acute respiratory failure
* infection (without septic shock)
* acute rheumatic disorder
* inflammatory bowel disease

Exclusion Criteria:

* patients with venous thromboembolism (VTE)
* active bleeding or at high risk of bleeding
* unable to take oral medication
* with diseases requiring ongoing treatment with anticoagulants or antiplatelets other than aspirin at a dose ≤ 165 mg/day.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6758 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (239):
- United States (47):
  - University Of Alabama At Birmingham Hospital, Birmingham, Alabama
  - Heart Center Research, Llc, Huntsville, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - Az Pulmonary Specialists Ltd, Scottsdale, Arizona
  - Fort Smith Lung Center, Fort Smith, Arkansas
  - Scripps Clinic/Scripps Health And Green Hospital, La Jolla, California
  - Va Long Beach Healthcare System, Long Beach, California
  - Univ. Of Southern Calif. /Norris Comprehensive Cancer Center, Los Angeles, California
  - Dr. Felt Medical Office, Oakland, California
  - Stanford University, Stanford, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Florida Hospital Celebration Health, Celebration, Florida
  - Research Alliance, Inc., Clearwater, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Pensacola Lung Group, Pensacola, Florida
  - Indian River Med. Ctr., Vero Beach, Florida
  - Atlanta Institute For Medical Research, Inc, Atlanta, Georgia
  - Pulmonary & Critical Care Of Atlanta, Atlanta, Georgia
  - Idaho Falls Infectious Diseases, Pllc, Idaho Falls, Idaho
  - West Suburban Hospital, Oak Park, Illinois
  - Infectious Disease Of Indiana Psc, Carmel, Indiana
  - Cotton-O-Neil Clinical Research Center, Topeka, Kansas
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Transplant Institute, Detriot, Michigan
  - University Of Missouri-Columbia, Columbia, Missouri
  - Mercury Street Medical Group, Pllc, Butte, Montana
  - Creighton University Medical Center, Omaha, Nebraska
  - Morristown Memorial Hospital, Mornstown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Staten Island University Hospital, Staten Island, New York
  - Mission Hospital, Inc, Asheville, North Carolina
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The Milton S Hershey Medical Center Of Penn. State Univ., Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Palmetto Nephrology Pa, Orangeburg, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Texas Health Presbyterian Dallas, Dallas, Texas
  - Michael E. De Bakey Veteran Affairs Medical Center, Houston, Texas
  - Sonterra Clinical Research, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University Of Utah Medical Center, Salt Lake City, Utah
  - Mcguire Va Medical Center, Richmond, Virginia
- Argentina (11):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Derqui-Pilar, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Munro, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (9):
  - Local Institution, Concord, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Woodville, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Ringwood East, Victoria
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Belgium (6):
  - Local Institution, Ottignies, Waals-Brabant
  - Local Institution, Antwerp
  - Local Institution, Brasschaat
  - Local Institution, Brussels
  - Local Institution, Huy
  - Local Institution, Leuven
- Brazil (7):
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (6):
  - Local Institution, Ajax, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Granby, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
- Chile (3):
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Rancagua, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
- Colombia (3):
  - Local Institution, Bogotá
  - Local Institution, Bucaramanga
  - Local Institution, Medellín
- Czechia (7):
  - Local Institution, Brno
  - Local Institution, Jindřichův Hradec
  - Local Institution, Kladno
  - Local Institution, Kyjov
  - Local Institution, Ostrava
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- Denmark (12):
  - Local Institution, Aalborg
  - Local Institution, Aarhus N
  - Local Institution, Arhus C
  - Local Institution, Frederiksberg
  - Local Institution, Glostrup Municipality
  - Local Institution, Hellerup
  - Local Institution, Herlev
  - Local Institution, Herning
  - Local Institution, Hvidovre
  - Local Institution, Odense
  - Local Institution, Randers NØ
  - Local Institution, Silkeborg
- France (10):
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Nancy
  - Local Institution, Nîmes
  - Local Institution, Paris
  - Local Institution, Saint-Etienne
  - Local Institution, Vernon
- Germany (10):
  - Local Institution, Bonn
  - Local Institution, Coburg
  - Local Institution, Darmstadt
  - Local Institution, Dresden
  - Local Institution, Hanover
  - Local Institution, Karlsbad
  - Local Institution, Lübeck
  - Local Institution, Mannheim
  - Local Institution, Offenbach
  - Local Institution, Witten
- Local Institution, Shatin, N.T., Hong Kong
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Dunaújváros
  - Local Institution, Eger
- India (16):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Visakhapatnam, Andhra Pradesh
  - Local Institution, Ahemdabad, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Indore, Madhya Pardesh
  - Local Institution, Pune, Maharashtra
  - Local Institution, Ludhiana, Punjab
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Coimbatore, Tamil Nadu
  - Local Institution, Madurai, Tamil Nadu
  - Local Institution, Noida, Uttar Pradesh
  - Local Institution, Ahmedabad
  - Local Institution, Bangalore
  - Local Institution, Hyderabad
  - Local Institution, Mumbai
  - Local Institution, New Delhi
- Israel (9):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
  - Local Institution, Ẕerifin
- Italy (7):
  - Local Institution, Chieti Scalo
  - Local Institution, Cremona
  - Local Institution, Padua
  - Local Institution, Piacenza
  - Local Institution, Reggio Emilia
  - Local Institution, Treviso
  - Local Institution, Vicenza
- Malaysia (3):
  - Local Institution, Kubang Kerian, Kelantan
  - Local Institution, Batu Caves, Selangor
  - Local Institution, Johor Bahru
- Mexico (6):
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Xalapa, Veracruz
  - Local Institution, Mérida, Yucatán
- Local Institution, Den Helder, Netherlands
- Local Institution, Kongsvinger, Norway
- Peru (4):
  - Local Institution, Lima, Lima Province
  - Local Institution, La Victoria, Lima region
  - Local Institution, Callao, Provincia Constitucional del Callao
  - Local Institution, Arequipa
- Philippines (3):
  - Local Institution, Cagayan de Oro, Misamis Oriental
  - Local Institution, Las Piñas
  - Local Institution, Quezon City
- Poland (9):
  - Local Institution, Bydgoszcz
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Nowa Sól
  - Local Institution, Poznan
  - Local Institution, Skierniewice
  - Local Institution, Warsaw
  - Local Institution, Wejherowo
  - Local Institution, Zielona Góra
- Russia (6):
  - Local Institution, Moscow
  - Local Institution, Odintsovo
  - Local Institution, Podolsk
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
- Local Institution, Singapore, Singapore
- South Africa (6):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, eManzimtoti, KwaZulu-Natal
  - Local Institution, Bellville, Western Cape
  - Local Institution, Groenkloof
- South Korea (4):
  - Local Institution, Guri-si, Gyeonggi-do
  - Local Institution, Seongnam-si, Gyeonggi-do
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (6):
  - Local Institution, Torrevieja, Alicante
  - Local Institution, Alcorcon(Madrid)
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville
  - Local Institution, Tarragona
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Lund
- Taiwan (2):
  - Local Institution, Yung-Kang City, Tainan
  - Local Institution, Taichung
- Turkey (Türkiye) (3):
  - Local Institution, Istanbul, Capa
  - Local Institution, Ankara, Dikimevi
  - Local Institution, Istanbul
- Ukraine (7):
  - Local Institution, Donetsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Lutsk
  - Local Institution, Lviv
  - Local Institution, Uzhhorod
  - Local Institution, Vinnitsa
- United Kingdom (5):
  - Local Institution, London, Greater London
  - Local Institution, Uxbridge, Middlesex
  - Local Institution, Newcastle, Tyne and Wear
  - Local Institution, Dudley, West Midlands
  - Local Institution, Hull, Yorkshire

REFERENCES:
- [Derived] Chi G, Goldhaber SZ, Kittelson JM, Turpie AGG, Hernandez AF, Hull RD, Gold A, Curnutte JT, Cohen AT, Harrington RA, Gibson CM. Effect of extended-duration thromboprophylaxis on venous thromboembolism and major bleeding among acutely ill hospitalized medical patients: a bivariate analysis. J Thromb Haemost. 2017 Oct;15(10):1913-1922. doi: 10.1111/jth.13783. Epub 2017 Sep 4. PMID 28762617
- [Derived] Marszalek J, Mehrsefat S, Chi G. The risk of stroke among acutely ill hospitalized medical patients: lessons from recent trials on extended-duration thromboprophylaxis. Expert Rev Hematol. 2017 Aug;10(8):679-684. doi: 10.1080/17474086.2017.1343662. Epub 2017 Jun 21. PMID 28617144
- [Derived] Sharma A, Chatterjee S, Lichstein E, Mukherjee D. Extended thromboprophylaxis for medically ill patients with decreased mobility: does it improve outcomes? J Thromb Haemost. 2012 Oct;10(10):2053-60. doi: 10.1111/j.1538-7836.2012.04874.x. PMID 22863355
- [Derived] Goldhaber SZ, Leizorovicz A, Kakkar AK, Haas SK, Merli G, Knabb RM, Weitz JI; ADOPT Trial Investigators. Apixaban versus enoxaparin for thromboprophylaxis in medically ill patients. N Engl J Med. 2011 Dec 8;365(23):2167-77. doi: 10.1056/NEJMoa1110899. Epub 2011 Nov 13. PMID 22077144
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient, first visit was June 2007 and last patient, last visit was May 2011. Acutely ill patients who had been hospitalized and had an expected hospitalization of an additional 3 or more days after randomization were enrolled.
Pre-assignment Details: 6758 enrolled; 6528 randomized to treatment. Reasons for non-randomization: 2 Adverse event (AE); 34 withdrew consent; 1 death; 3 poor/non-compliance; 162 no longer met study criteria; 2 administrative reason by Sponsor; 26 other reasons.
Groups:
- Apixaban 2.5 mg Oral: Oral administration of 2.5 mg apixaban tablets twice daily (BID) for 30 days plus placebo matching enoxaparin 40 mg QD while in hospital and for a minimum of 6 days.
- Enoxaparin 40 mg Subcutaneous: Subcutaneous (SC) administration of 40 mg enoxaparin once daily (QD) for a minimum of 6 days plus placebo tablets matching apixaban 2.5 mg for 30 days.
Period: Overall Study
Arm/Group | Apixaban 2.5 mg Oral | Enoxaparin 40 mg Subcutaneous
Started | 3255 | 3273
Completed | 2442 | 2516
Not Completed | 813 | 757
Not completed — Death | 40 | 47
Not completed — Adverse Event | 284 | 260
Not completed — Withdrawal by Subject | 299 | 271
Not completed — Lost to Follow-up | 72 | 71
Not completed — Poor/Non-compliance | 46 | 33
Not completed — No longer met criteria | 41 | 37
Not completed — Administrative reason by Sponsor | 1 | 0
Not completed — non-specified | 29 | 38
Not completed — treated for 1 day; missing status/reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Participants
Groups:
- Apixaban 2.5 mg: Oral administration of 2.5 mg apixaban tablets twice daily (BID) for 30 days plus placebo matching enoxaparin 40 mg QD while in hospital and for a minimum of 6 days.
- Enoxaparin 40 mg: Subcutaneous (SC) administration of 40 mg enoxaparin once daily (QD) for a minimum of 6 days plus placebo tablets matching apixaban 2.5 mg for 30 days.
- Total: Total of all reporting groups
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg | Total
Number analyzed (Participants) | 3255 | 3273 | 6528
Age, Continuous [Median (Full Range); unit: years] | 68.0 [40 to 101] | 67.0 [40 to 98] | 67.0 [40 to 101]
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 1401 | 1411 | 2812
  Greater than, equal to (>=) 65 and < 75 years | 890 | 884 | 1774
  >= 75 years | 964 | 978 | 1942
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1629 | 1696 | 3325
  Male | 1626 | 1577 | 3203
Region of Enrollment [Number; unit: participants] — Randomized Participants.
  participants
    United States | 625 | 620 | 1245
    Philippines | 22 | 22 | 44
    Hong Kong | 26 | 26 | 52
    Taiwan | 8 | 7 | 15
    Spain | 51 | 50 | 101
    Ukraine | 270 | 276 | 546
    Chile | 65 | 65 | 130
    Israel | 168 | 168 | 336
    Russian Federation | 632 | 632 | 1264
    Colombia | 10 | 14 | 24
    Italy | 35 | 34 | 69
    India | 198 | 202 | 400
    France | 203 | 200 | 403
    Malaysia | 9 | 11 | 20
    Denmark | 49 | 54 | 103
    Australia | 51 | 49 | 100
    Peru | 119 | 121 | 240
    South Africa | 52 | 48 | 100
    Netherlands | 1 | 0 | 1
    Korea, Republic of | 33 | 33 | 66
    Turkey | 9 | 10 | 19
    Austria | 5 | 7 | 12
    United Kingdom | 195 | 194 | 389
    Hungary | 18 | 16 | 34
    Czech Republic | 53 | 56 | 109
    Mexico | 58 | 59 | 117
    Canada | 45 | 47 | 92
    Argentina | 78 | 77 | 155
    Brazil | 41 | 45 | 86
    Belgium | 21 | 22 | 43
    Poland | 57 | 60 | 117
    Singapore | 8 | 12 | 20
    Norway | 3 | 2 | 5
    Germany | 35 | 32 | 67
    Sweden | 2 | 2 | 4
Participants with Risk Factors [Number; unit: participants] — This baseline measures randomized participants.
  participants
    Previous Venous Thromboembolism (VTE) | 141 | 124 | 265
    Estrogenic Hormone Therapy | 49 | 27 | 76
    History of Malignancy | 312 | 320 | 632
    Chronic Heart Failure | 1531 | 1537 | 3068

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Composite of Adjudicated Total Venous Thromboembolism (VTE) and VTE-related Death During the Intended Treatment Period - Primary Efficacy Population
Description: VTE: nonfatal pulmonary embolism (PE), symptomatic deep vein thrombosis (DVT), or asymptomatic proximal DVT detected by ultrasound. VTE-related death: fatal PE or sudden death for which VTE could not be excluded as a cause. Intended Treatment Period=period that started on day of randomization: period ended (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; period ended (for not treated) 32 days after randomization. A bilateral compression ultrasound (CUS) was performed between Days 5 and 14 for detection of asymptomatic proximal DVT unless a symptomatic VTE was confirmed prior. CUS was also performed on Day 30 ± 2 except for those participants who had a confirmed symptomatic VTE or proximal asymptomatic DVT prior to that time. All efficacy events were adjudicated by the Independent Central Adjudication Committee (ICAC). Event rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: Those randomized (without suspected VTE) who had an adjudicated and evaluable ultrasound at end of intended treatment; or (with suspected VTE) had VTE events adjudicated as non-events and had an adjudicated and evaluable ultrasound at end of intended treatment, or had an adjudicated total VTE-related death.
Measure: Number (95% Confidence Interval); unit: Event rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2211 | 2284
Event rate (%) | 2.71 [2.11 to 3.49] | 3.06 [2.43 to 3.86]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; To conclude superiority of apixaban versus enoxaparin on the primary efficacy endpoint, the upper bound of the two-sided 95.004% confidence interval (CI) for the relative risk (pa/ pe) must be less than 1; Test type: Superiority or Other; p = 0.4364, Mantel Haenszel; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.62 to 1.23]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.39, 95% CI 2-sided [-1.37 to 0.59]

2. Secondary Outcome: Incidence of Adjudicated Total VTE and VTE-Related Death During Parenteral Treatment in Key Secondary Efficacy Evaluable Participants
Description: Parenteral study drug=active or placebo enoxaparin. Parenteral treatment: started on the first dose of parenteral study drug and ended the day after the last dose of parenteral study drug. Key Secondary Efficacy population: all who received at least 1 dose of parenteral study drug and: (those without suspected VTE events during Parenteral Treatment) had an adjudicated evaluable ultrasound performed at the end of Parenteral Treatment; or (those with suspected VTE events during Parenteral Treatment) had those suspected VTE events adjudicated as non-events, and had an adjudicated evaluable ultrasound performed at the end of Parenteral Treatment; or had an adjudicated total VTE during Parenteral Treatment; or had an adjudicated VTE-related death during Parenteral Treatment. Event rate (%): n/N*100 (n=number with observation; N=total secondary efficacy evaluable participants).
Time Frame: Day 1 to last dose of parenteral study drug plus 1 day
Population: Those randomized (without suspected VTE) who had an adjudicated and evaluable ultrasound at end of parenteral treatment; or (with suspected VTE) had VTE events adjudicated as non-events and had adjudicated and evaluable ultrasound at end of parenteral treatment, or had an adjudicated VTE-related death during the Parenteral Treatment Period.
Measure: Number (95% Confidence Interval); unit: Event rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2485 | 2488
Event rate (%) | 1.73 [1.28 to 2.33] | 1.61 [1.18 to 2.19]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Formal testing of noninferiority for the key secondary efficacy endpoint was not performed since the superiority of the primary efficacy endpoint was not demonstrated; Test type: Superiority or Other; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.69 to 1.63]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = 0.10, 95% CI 2-sided [-0.61 to 0.81]

3. Secondary Outcome: Incidence of Adjudicated Total VTE and VTE-Related Death During Parenteral Treatment in Secondary Efficacy Evaluable Participants
Description: Parenteral study drug=active or placebo enoxaparin. Parenteral treatment: started on the first dose of parenteral study drug and ended the day after the last dose of parenteral study drug. Secondary Efficacy Evaluable includes those who had an adjudicated, evaluable ultrasound at end of parenteral treatment and for those with a suspected symptomatic event, the result of the adjudication for the symptomatic event was not inadequate; or those with an adjudicated event that was part of the composite endpoint.. Event rate (%): n/N*100 (n=number with observation; N=total secondary efficacy evaluable participants).
Time Frame: Day 1 to last dose of parenteral study drug plus 1 day
Population: Secondary Efficacy Evaluable includes those who have an adjudicated, evaluable ultrasound at end of parenteral treatment and for those with a suspected symptomatic event, the result of the adjudication for the symptomatic event is not inadequate; or those with an adjudicated event that is part of the composite endpoint.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2344 | 2380
Event Rate (%) | 1.66 [1.22 to 2.28] | 1.51 [1.09 to 2.10]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.70 to 1.71]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = 0.14, 95% CI 2-sided [-0.57 to 0.85]

4. Secondary Outcome: Incidence of Adjudicated Total VTE or All-Cause Death With Onset During the Intended Treatment Period
Description: Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. VTE: nonfatal (N-F) PE, symptomatic DVT, or asymptomatic proximal DVT detected by ultrasound. VTE-related death: fatal PE or sudden death for which VTE cannot be excluded as a cause. All-Cause Death (A-C Death). Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: Those randomized with adjudicated and evaluable ultrasound at the end of the intended treatment period; for those with a suspected symptomatic event, the adjudication result was not inadequate; includes all those randomized who have an adjudicated event associated with the endpoint during Intended Treatment.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2297 | 2369
Event Rate (%) | 6.44 [5.51 to 7.53] | 6.63 [5.69 to 7.71]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.78 to 1.20]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.24, 95% CI 2-sided [-1.65 to 1.17]

5. Secondary Outcome: Incidence of Adjudicated Proximal DVT, Non-Fatal PE or All-Cause Death With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2297 | 2368
Event Rate (%) | 6.44 [5.51 to 7.53] | 6.50 [5.58 to 7.58]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.79 to 1.22]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.12, 95% CI 2-sided [-1.52 to 1.29]

6. Secondary Outcome: Incidence of Adjudicated Proximal DVT, Non-Fatal PE or VTE-Related Death, With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. VTE-related death: fatal PE or sudden death for which VTE cannot be excluded as a cause. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2211 | 2283
Event Rate (%) | 2.71 [2.11 to 3.49] | 2.93 [2.32 to 3.72]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.65 to 1.29]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.26, 95% CI 2-sided [-1.23 to 0.71]

7. Secondary Outcome: Incidence of Adjudicated VTE-Related Death With Onset During the Intended Treatment Period in Randomized Participants
Description: as for outcome 6
Time Frame: Intended Treatment Period
Population: All Randomized Participants.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3255 | 3273
Event Rate (%) | 0.06 [0.00 to 0.24] | 0.09 [0.02 to 0.29]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.11 to 4.05]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.03, 95% CI 2-sided [-0.16 to 0.10]

8. Secondary Outcome: Incidence of Adjudicated Symptomatic VTE or All-Cause Death With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. VTE: nonfatal PE, symptomatic DVT, or asymptomatic proximal DVT detected by ultrasound. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: Randomized participants except those with an inadequate assessment for symptomatic events that are part of the endpoint during the intended treatment were analyzed.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3251 | 3269
Event Rate (%) | 3.11 [2.56 to 3.77] | 3.46 [2.88 to 4.14]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.68 to 1.16]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.38, 95% CI 2-sided [-1.25 to 0.48]

9. Secondary Outcome: Symptomatic Adjudicated VTE or VTE-Related Death With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. VTE: nonfatal PE, symptomatic DVT, or asymptomatic proximal DVT detected by ultrasound. VTE-related death: fatal PE or sudden death for which VTE cannot be excluded as a cause. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3251 | 3266
Event Rate (%) | 0.40 [0.23 to 0.69] | 0.80 [0.54 to 1.17]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.26 to 0.96]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.40, 95% CI 2-sided [-0.78 to -0.03]

10. Secondary Outcome: Incidence of All VTE or Major Bleeding or All-Cause Death During the Intended Treatment Period
Description: as for outcome 9
Time Frame: Intended Treatment Period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2304 | 2371
Event Rate (%) | 7.16 [6.18 to 8.29] | 6.83 [5.88 to 7.93]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.84 to 1.28]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = 0.28, 95% CI 2-sided [-1.18 to 1.73]

11. Secondary Outcome: Incidence of Adjudicated PE With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. PE: non-fatal or fatal. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3251 | 3266
Event Rate (%) | 0.22 [0.10 to 0.46] | 0.24 [0.12 to 0.50]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.32 to 2.43]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.03, 95% CI 2-sided [-0.26 to 0.20]

12. Secondary Outcome: Incidence of Adjudicated Non-Fatal PE With Onset During the Intended Treatment Period
Description: as for outcome 5
Time Frame: Intended Treatment Period
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3251 | 3266
Event Rate (%) | 0.22 [0.10 to 0.46] | 0.24 [0.12 to 0.50]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.32 to 2.43]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.03, 95% CI 2-sided [-0.26 to 0.20]

13. Secondary Outcome: Incidence of Adjudicated Symptomatic DVT With Onset During the Intended Treatment Period
Description: as for outcome 5
Time Frame: Intended Treatment Period
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3255 | 3273
Event Rate (%) | 0.15 [0.06 to 0.37] | 0.49 [0.30 to 0.80]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.31, 95% CI 2-sided [0.11 to 0.83]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.34, 95% CI 2-sided [-0.62 to -0.07]

14. Secondary Outcome: Incidence of Adjudicated Proximal DVT With Onset During the Intended Treatment Period
Description: Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. A bilateral compression ultrasound (CUS) was performed between Days 5 and 14 for detection of asymptomatic proximal DVT unless a symptomatic VTE was confirmed prior. CUS was also performed on Day 30 ± 2 except for those participants who had a confirmed symptomatic VTE or proximal asymptomatic DVT prior to that time. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2207 | 2276
Event Rate (%) | 2.40 [1.84 to 3.14] | 2.50 [1.94 to 3.24]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.65 to 1.37]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.14, 95% CI 2-sided [-1.04 to 0.76]

15. Secondary Outcome: Incidence of Adjudicated Symptomatic Distal DVT With Onset During the Intended Treatment Period
Description: Events were adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: Randomized participants, except those with an inadequate assessment for symptomatic events that are part of the endpoint during the intended treatment period, were analyzed.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3255 | 3273
Event Rate (%) | 0.00 [0.00 to 0.15] | 0.15 [0.06 to 0.37]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Note: Relative risk was not estimable (0.0); only risk difference could be estimated; Test type: Superiority or Other; Risk Difference (RD) = -0.15, 95% CI 2-sided [-0.29 to -0.02]

16. Secondary Outcome: Incidence of Adjudicated Symptomatic Proximal DVT With Onset During the Intended Treatment Period
Description: as for outcome 14
Time Frame: Intended Treatment Period
Population: Randomized participants, except those with an inadequate assessment for symptomatic events that are part of the endpoint during the intended treatment, were analyzed.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3255 | 3273
Event Rate (%) | 0.15 [0.06 to 0.37] | 0.37 [0.20 to 0.65]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 0.41, 95% CI 2-sided [0.14 to 1.16]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.22, 95% CI 2-sided [-0.47 to 0.03]

17. Primary Outcome: Incidence of Major Bleeding During the Treatment Period in Treated Participants
Description: Major bleeding was adjudicated by an ICAC using criteria from the International Society on Thrombosis and Hemostasis (ISTH) and was defined as acute clinically overt bleeding: associated with a fall in hemoglobin of 2 grams per deciliter (g/dL) or more, or leading to a transfusion of 2 or more units of packed red blood cells or 1000 milliliters (mL) or more of whole blood, or bleeding in a critical site or bleeding which is fatal. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Day 1, first dose of study drug, to last dose of study drug plus 2 days
Population: Participants who received at least one dose of study drug were analyzed (As Treated population). Participants were categorized to the group to which they were randomized, unless the same incorrect treatment was received throughout the study; in such case, the As Treated were equal to the treatment received.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
Event Rate (%) | 0.47 [0.28 to 0.79] | 0.19 [0.08 to 0.42]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Adjusted difference of event rates takes the stratification factor into consideration: previous VTE (yes, no) and active or previous cancer (yes, no); Test type: Superiority or Other; p = 0.0437, Mantel Haenszel — The Mantel-Haenszel test stratified by the stratification factors will be used at the one-sided alpha=0.025 level; Adjusted Difference of event rates = 0.29, 95% CI 2-sided [0.01 to 0.57]

18. Primary Outcome: Incidence of Clinically Relevant Non-Major (CRNM) Bleeding During the Treatment Period in Treated Participants
Description: Bleeding was adjudicated by an ICAC using criteria from the ISTH. CRNM bleeding: acute clinically overt bleeding compromising hemodynamics; leading to hospitalization; traumatic subcutaneous hematoma; intramuscular hematoma; epistaxis that lasted for more than 5 minutes, was repetitive or led to an intervention; spontaneous gingival bleeding; spontaneous hematuria; macroscopic gastrointestinal hemorrhage (including at least 1 episode of melena or hematemesis, if clinically apparent with positive results on a fecal occult-blood test); rectal blood loss. Treatment Period=includes measurements or events with onset from first dose of study drug through 2 days after the last dose of study drugs for bleeding endpoints. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Day 1, first dose of study drug, to last dose of study drug plus 2 days
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Event Rate (%):
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
Event Rate (%): | 2.26 [1.80 to 2.84] | 1.90 [1.48 to 2.43]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Adjusted Difference of event rates = 0.36, 95% CI 2-sided [-0.33 to 1.06]

19. Primary Outcome: Incidence of Composite of Major or Clinically Relevant Non-Major (CRNM) Bleeding During the Treatment Period in Treated Participants
Description: Bleeding was adjudicated by an ICAC using criteria from the ISTH. Major bleeding: acute clinically overt bleeding: associated with a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of 2 or more units of packed red blood cells or 1000 mL or more of whole blood, or bleeding in a critical site or bleeding which is fatal. CRNM bleeding: acute clinically overt bleeding compromising hemodynamics; leading to hospitalization; traumatic subcutaneous hematoma; intramuscular hematoma; epistaxis that lasted for more than 5 minutes, was repetitive or led to an intervention; spontaneous gingival bleeding; spontaneous hematuria; macroscopic gastrointestinal hemorrhage; rectal blood loss. Treatment Period=onset from first dose of study drug through 2 days after last dose of study drugs. Incidence: Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Day 1, first dose of study drug, to last dose of study drug plus 2 days
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
Event Rate (%) | 2.67 [2.16 to 3.29] | 2.08 [1.64 to 2.64]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Adjustted difference of event rates = 0.59, 95% CI 2-sided [-016 to 1.33]

20. Primary Outcome: Incidence of All Bleeding During the Treatment Period in Treated Participants
Description: Bleeding was adjudicated by an ICAC using criteria from the ISTH. Treatment Period=includes measurements or events with onset from first dose of study drug through 2 days after the last dose of study drugs, for bleeding endpoints. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Day 1, first dose of drug to last dose of drug plus 2 days
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
Event Rate (%) | 7.73 [6.85 to 8.71] | 6.81 [5.99 to 7.73]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Adjusted Difference of Event Rates = 0.87, 95% CI 2-sided [-0.40 to 2.14]

21. Secondary Outcome: Incidence of Adjudicated Asymptomatic Proximal DVT With Onset During the Intended Treatment Period
Description: A bilateral compression ultrasound (CUS) was performed between Days 5 and 14 for detection of asymptomatic proximal DVT unless a symptomatic VTE was confirmed prior. CUS was also performed on Day 30 ± 2 except for those participants who had a confirmed symptomatic VTE or proximal asymptomatic DVT prior to that time. Events adjudicated by ICAC. Intended Treatment Period=period that starts on day of randomization: period ends (for treated) at latter of a) 2 days after last dose of study drug and b) 32 days after first dose of study drug; (for not treated) period ends 32 days after randomization. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants).
Time Frame: Intended Treatment Period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2206 | 2269
Event Rate (%) | 2.36 [1.80 to 3.09] | 2.12 [1.60 to 2.80]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.74 to 1.61]
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Test type: Superiority or Other; Risk Difference (RD) = 0.20, 95% CI 2-sided [-0.66 to 1.07]

22. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Bleeding AEs, Deaths, and Discontinuations Due to AEs During the Treatment Period in Treated Participants
Description: Treatment Period=includes measurements or events with onset from first dose of study drug through 2 days after the last dose of study drugs for AEs, and 30 days after last dose of study drugs for SAEs and deaths.
Time Frame: Day 1, first dose of study drug, to last dose of study drug plus 2 days (AEs), plus 30 days (SAEs, Deaths)
Population: Participants who received at least one dose of study drug were analyzed (As Treated population).
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
participants
  AEs | 1871 | 1910
  SAEs | 611 | 601
  Bleeding AEs | 244 | 221
  Discontinuations Due to AE | 290 | 262
  Deaths | 131 | 133

23. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure in Treated Participants During Treatment Period
Description: Diastolic blood pressure was obtained during Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days. Blood pressure was measured in millimeters of mercury (mmHg) and could have been taken with the participant either sitting, standing, or supine.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: Participants who received at least one dose of study drug, had a baseline value, and had a value on the day specified were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2227 | 2301
mmHg
  Day of Discharge from Hospital (N=1607, 1625) | -1.0 (12.69) | -0.4 (12.32)
  Day 30 of Treatment + 2 (N=2227,2301) | 0.0 (12.91) | -0.5 (12.78)

24. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure in Treated Participants During Treatment Period
Description: Systolic blood pressure was obtained during Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days. Blood pressure was measured in millimeters of mercury (mmHg) and could have been taken either sitting, standing, or supine.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2227 | 2301
mmHg
  Discharge from Hospital (N=1607, 1625) | -3.0 (19.12) | -2.4 (19.80)
  Day 30 of Treatment + 2 (N=2227, 2301) | -2.3 (19.79) | -2.9 (20.61)

25. Secondary Outcome: Mean Change From Baseline in Heart Rate in Treated Participants
Description: Heart Rate was obtained during Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days. Heart rate was measured in beats per minute (bpm) and could have been taken with participants either sitting, standing, or supine.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2225 | 2299
bpm
  Hospital Discharge (N=1606,1622) | -5.4 (14.08) | -5.1 (14.07)
  Day 30 of treatment (N=2225,2299) | -4.0 (15.62) | -4.3 (14.83)

26. Secondary Outcome: Number of Participants With Marked Abnormalities in Hematology Laboratory Tests During Treatment Period in Treated Participants
Description: Lower limit of normal (LLN). Upper limit of normal (ULN). Pre-therapy (PreRx). Absolute (Abs) neutrophil count, bands + neutrophils (ANC). Cells per microliter (c/µL). Grams per deciliter (g/dL). Cells per Liter (c/L). Millimeter (MM). Absolute (Abs). Hemoglobin: >2 g/dL decrease compared to PreRx value or value <=8 g/dL; Hematocrit: <0.75*PreRx; Erythrocytes: <0.75*PreRx c/µL; Leukocytes: <0.75*LLN or > 1.25*ULN, if PreRx <LLN then use <0.8*PreRx or >ULN, if PreRx >ULN then use >1.2*PreRx or < LLN; Platelet count: < 100*10^9 c/L; ANC: < 1.00*10^3 c/µL; Abs eosinophils: > 0.75*10^3 c/µL; Abs Basophils: > 400/MM^3; Abs Monocytes > 2000/MM^3; Abs Lymphocytes: < 0.750*10*3 c/ µL or > 7.5*10^3 c/ µL. Samples were obtained at Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: Participants who received at least one dose of study drug, had a pre-therapy value, and had a value on the day specified were analyzed.
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2835 | 2871
participants
  Hemoglobin >2 g/dL decrease (N=2835, 2871) | 133 | 98
  Hematocrit <0.75*PreRx (N=2688, 2722) | 23 | 17
  Platelet Count < 100*10^9 c/L (N=2761, 2799) | 9 | 7
  Erythrocytes <0.75*PreRx c/µL (N=2697, 2730) | 28 | 16
  Leukocytes <0.75*LLN (N= 2835, 2869) | 64 | 55
  Leukocytes > 1.25*ULN (N=2835, 2869) | 331 | 283
  Abs Eosinophils > 0.75*10^3 c/µL (N=20, 24) | 1 | 1
  Abs Lymphocytes < 0.750*10*3 c/ µL (N=20, 24) | 4 | 2
  Abs Monocytes > 2000/MM^3 (N= 19, 25) | 1 | 0

27. Secondary Outcome: Number of Participants With Marked Abnormalities in Electrolyte Laboratory Tests During Treatment Period in Treated Participants
Description: Bicarbonate milliequivalents/Liter (mEq/L) Low/High: < 0.75*LLN or > 1.25*ULN, or if PreRx < LLN then use < 0.75* PreRx or > ULN if PreRx > ULN then use > 1.25*PreRx or < LLN; Serum Calcium mg/dL Low/High: < 0.8*LLN or > 1.2*ULN, or if PreRx < LLN then use < 0.75*PreRx or > ULN if PreRx > ULN then use > 1.25*PreRx or < LLN; Serum Chloride mEq/L: < 0.9*LLN or > 1.1*ULN, or if PreRx < LLN then use < 0.9*PreRx or > ULN if PreRx > ULN then use > 1.1*PreRx or < LLN; Serum Potassium mEq/L: < 0.9*LLN or > 1.1*ULN, or if PreRx < LLN then use < 0.9*PreRx or > ULN if PreRx > ULN then use > 1.1*PreRx or < LLN; Serum Sodium mEq/L: < 0.95*LLN or > 1.05*ULN, or if PreRx < LLN then use < 0.95*PreRx or > ULN if PreRx > ULN then use > 1.05*PreRx or < LLN. Samples obtained at Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2862 | 2893
participants
  Calcium < 0.8*LLN (N=2861, 2893) | 6 | 8
  Calcium > 1.2*ULN (N=2861, 2893) | 3 | 3
  Chloride < 0.9*LLN (N=2861, 2886) | 25 | 25
  Chloride > 1.1*ULN (N=2861, 2886) | 5 | 1
  Bicarbonate < 0.75*LLN (N=2831, 2855) | 5 | 6
  Bicarbonate > 1.25*ULN (N=2831, 2855) | 6 | 4
  Potassium < 0.9*LLN (N=2851, 2878) | 61 | 58
  Potassium > 1.1*ULN (N=2851, 2878) | 140 | 137
  Sodium < 0.95*LLN (N=2862, 2888) | 23 | 25
  Sodium > 1.05*ULN (N=2862, 2888) | 9 | 6

28. Secondary Outcome: Number of Participants With Marked Abnormalities in Kidney and Liver Function Laboratory Tests During the Treatment Period in Treated Participants
Description: Blood urea nitrogen (BUN), milligrams/deciliter (mg/dL), units per liter (U/L). BUN mg/dL > 1.5*ULN; Creatinine mg/dL: > 1.5*ULN; Alanine aminotransferase (ALT) U/L: > 3*ULN; Aspartate aminotransferase (AST) U/L: > 3*ULN; Alkaline phosphatase U/L: > 2*ULN; Bilirubin Direct mg/dL: > 1.5*ULN; Bilirubin Total mg/dL: > 2*ULN. Samples for laboratories obtained at Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) plus 2 days.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2866 | 2895
participants
  Alkaline phosphatase U/L > 2*ULN(N=2866, 2895) | 35 | 47
  ALT U/L > 3*ULN (N=2827, 2861) | 23 | 33
  AST U/L > 3*ULN (N=2831, 2863) | 24 | 29
  Bilirubin Direct mg/dL > 1.5*ULN (N=2782, 2821) | 123 | 106
  Bilirubin Total mg/dL > 2*ULN (N=2853, 2884) | 17 | 15
  BUN mg/dL > 1.5*ULN (N=2864, 2891) | 194 | 188
  Creatinine mg/dL > 1.5*ULN (N=2862, 2892) | 150 | 156

29. Secondary Outcome: Number of Participants With Marked Abnormalities in Glucose, Creatine Kinase, Uric Acid, and Total Protein Laboratory Tests During the Treatment Period in Treated Participants
Description: Creatine kinase High: >5*ULN Units/Liter (U/L); Total Protein High/Low: < 0.9 *LLN or > 1.1*ULN, or if PreRx < LLN then use 0.9* PreRx or > ULN if PreRx > ULN then use 1.1 *PreRx or <LLN; Uric acid High: > 1.5* ULN, or if PreRx > ULN then use > 2 *PreRx. Glucose Fasting: <0.9*LLN or > 1.5*ULN or if PreRx < LLN then use < 0.8*PreRx or > ULN, if PreRx > ULN then use >2.0*PreRx. Samples obtained at Screening/Enrollment Visit (Day 1, prior to drug being administered), on the day of hospital discharge, Day 30 (last day of treatment) ± 2days.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2864 | 2890
participants
  Glucose Fasting <0.9*LLN (N=284,287) | 5 | 3
  Glucose Fasting > 1.5*ULN (N=284,287) | 39 | 30
  Total Protein < 0.9 *LLN (N=2864, 2890) | 78 | 51
  Total Protein > 1.1*ULN (N=2864, 2890) | 16 | 8
  Creatine kinase >5*ULN U/L(N=2856, 2888) | 8 | 10
  Uric acid > 1.5* ULN (N=2862, 2889) | 47 | 44

30. Secondary Outcome: Incidence of Events of Special Interest of Adjudicated Myocardial Infarction, Stroke, and Thrombocytopenia During the Treatment Period in Treated Participants
Description: Events of Special Interest include: adjudicated thrombocytopenia, adjudicated myocardial infarction (MI), adjudicated stroke, and adjudicated MI or stroke. Incidence determined by Event Rate (%): n/N*100 (n=number with observation; N=total efficacy evaluable participants). Treatment Period includes measurements or events with onset from first dose of study drug through 2 days after the last dose of study drugs.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: MI and thrombocytopenia categories: participants who received at least one dose of study drug. MI or stroke category: treated participants except those who did not have MI and had an inadequate assessment for stroke. Stroke category: treated participants except those with an inadequate assessment for stroke during the treatment period.
Measure: Number (95% Confidence Interval); unit: Event Rate (%)
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
Event Rate (%)
  MI or stoke (N=3183, 3216) | 0.38 [0.21 to 0.67] | 0.37 [0.21 to 0.66]
  MI (N=3184, 3217) | 0.22 [0.10 to 0.47] | 0.12 [0.04 to 0.34]
  Stroke (N=3183, 3216) | 0.16 [0.06 to 0.38] | 0.25 [0.12 to 0.50]
  Thrombocytopenia (N=3184, 3217) | 0.19 [0.08 to 0.42] | 0.09 [0.02 to 0.29]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Adjusted difference in event rates in MI or stroke; Test type: Superiority or Other; Adjusted Event rate difference = -0.00, 95% CI 2-sided [-0.30 to 0.29] — stratification factor: previous VTE (yes, no), and active or previous cancer (yes, no)
Statistical Analysis 2: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Adjusted difference of event rates for myocardial infarction; Test type: Superiority or Other; Adjusted difference of event rates = 0.09, 95% CI 2-sided [-0.11 to 0.30] — stratification factor: previous VTE (yes, no), and active or previous cancer (yes, no)
Statistical Analysis 3: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Adjusted difference in event rates for stroke; Test type: Superiority or Other; Adjusted difference in event rates = -0.10, 95% CI 2-sided [-0.32 to 0.12]
Statistical Analysis 4: Comparison: Apixaban 2.5 mg vs Enoxaparin 40 mg; Adjusted difference of event rates in thrombocytopenia; Test type: Superiority or Other; Adjusted difference in event rates = 0.09, 95% CI 2-sided [-0.09 to 0.28] — stratification factor: previous VTE (yes, no), and active or previous cancer (yes, no)

31. Secondary Outcome: Number of Participants With Events of Special Interest for Liver Function and Neurology During Treatment Period in Treated Participants With Available Measurements
Description: Special interest include: liver function test increases, AEs related to liver function, and neurologic AEs. Treatment Period includes measurements or events with onset from first dose of study drug through 2 days after the last dose of study drug when summarizing AEs and through 30 days after the last dose when summarizing SAEs.
Time Frame: Day 1 to last dose of study drug plus 2 days (AEs) and plus 30 days (SAEs)
Population: Participants who received at least one dose of study drug, and had available laboratory results associated with the event and treatment group.
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 3184 | 3217
participants
  Neurologic AEs | 45 | 42
  Neurologic SAEs | 5 | 1
  Liver-related AEs | 127 | 142
  Liver-related SAEs | 9 | 12

32. Secondary Outcome: Number of Participants With Liver-Related Elevations During the Treatment Period in Treated Participants
Description: Liver function tests: Alanine aminotransferase (ALT) U/L; Aspartate aminotransferase (AST) U/L; Alkaline phosphatase U/L; Total Bilirubin (TBili) mg/dL. Elevations consist of >3*Upper Limit of Normal (ULN) for ALT and AST and elevation of >2*ULN for Bilirubin.
Time Frame: Day 1 to last dose of study drug plus 2 days
Population: Participants who received at least one dose of study drug and had available laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Enoxaparin 40 mg
Number analyzed (Participants) | 2853 | 2884
participants
  AST Elevation >3*ULN (N=2831, 2863) | 23 | 28
  ALT Elevation >3*ULN (N=2827, 2861) | 22 | 32
  AST + ALT >3*ULN on same date (N= 2827, 2861) | 14 | 13
  TBili >2*ULN (N= 2853, 2884) | 13 | 14
  ALT or AST >3*ULN + TBili >2*ULN (N=2818,2855) | 2 | 2
  ALT>3*ULN + TBili >2*ULN (N=2817, 2853) | 0 | 2

ADVERSE EVENTS:
Time Frame: Day 1, first dose of study drug, to last dose of study drug plus 2 days (AEs), plus 30 days (SAEs, Deaths).
Description: No AE met or exceeded the 5% frequency threshold. Participants who received at least one dose of study drug were analyzed.
Groups:
- Apix 2.5mg BID: Oral administration of 2.5 mg apixaban tablets twice daily (BID) for 30 days plus placebo matching enoxaparin 40 mg QD while in hospital and for a minimum of 6 days.
- Enox 40mg QD: Subcutaneous (SC) administration of 40 mg enoxaparin once daily (QD) for a minimum of 6 days plus placebo tablets matching apixaban 2.5 mg for 30 days.
Arm/Group | Apix 2.5mg BID | Enox 40mg QD
Serious Adverse Events (participants affected / at risk) | 611/3184 | 601/3217
Other Adverse Events (participants affected / at risk) | 0/3184 | 0/3217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apix 2.5mg BID (N=3184) | Enox 40mg QD (N=3217)
Anuria (Renal and urinary disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 19
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 8 | 7
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 3
Diabetic gangrene (Infections and infestations) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Gangrene (Infections and infestations) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Nasal abscess (Infections and infestations) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urine uric acid abnormal (Investigations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Angina pectoris (Cardiac disorders) | 1 | 2
Aortic valve disease mixed (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 14 | 15
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchitis (Infections and infestations) | 7 | 10
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bundle branch block left (Cardiac disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure (Cardiac disorders) | 50 | 28
Cardiomyopathy (Cardiac disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Congestive cardiomyopathy (Cardiac disorders) | 2 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 25 | 22
Depression (Psychiatric disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 2
Ischaemic ulcer (General disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Asthenia (General disorders) | 2 | 2
Bleeding varicose vein (Vascular disorders) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 6 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 91 | 103
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 9
Femoral artery occlusion (Vascular disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Headache (Nervous system disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Hypertensive crisis (Vascular disorders) | 0 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 10
Kidney infection (Infections and infestations) | 1 | 0
Liver function test abnormal (Investigations) | 2 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 0
Mycobacterium test positive (Investigations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 2
Pyrexia (General disorders) | 1 | 3
Renal failure chronic (Renal and urinary disorders) | 3 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 26 | 34
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 2
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 4 | 5
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Accelerated hypertension (Vascular disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 | 20
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 12 | 11
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Clonic convulsion (Nervous system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Distributive shock (Vascular disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Haemorrhage (Vascular disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia (Infections and infestations) | 54 | 40
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pyothorax (Infections and infestations) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Septic shock (Infections and infestations) | 6 | 6
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 4
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 2 | 5
Cardiac failure congestive (Cardiac disorders) | 31 | 32
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 2
Device related sepsis (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 4
Infected skin ulcer (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 8 | 13
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myasthenic syndrome (Nervous system disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 2
Radiculopathy (Nervous system disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 10 | 7
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sudden death (General disorders) | 4 | 6
Thrombosis (Vascular disorders) | 1 | 3
Troponin I increased (Investigations) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 4
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Angina unstable (Cardiac disorders) | 5 | 5
Ascites (Gastrointestinal disorders) | 0 | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 4 | 3
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Myocardial rupture (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Nephritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oedema peripheral (General disorders) | 4 | 2
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 2
Pain (General disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 12 | 12
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Sudden cardiac death (General disorders) | 2 | 3
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 3
Vitreous haemorrhage (Eye disorders) | 1 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 5 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 10 | 7
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Death (General disorders) | 6 | 10
Diverticulitis (Infections and infestations) | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 7 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hallucinations, mixed (Psychiatric disorders) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multi-organ failure (General disorders) | 5 | 1
Myeloid metaplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 9 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory tract infection (Infections and infestations) | 4 | 5
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Systemic candida (Infections and infestations) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 8 | 3
Aortic stenosis (Vascular disorders) | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 4 | 3
Bacteraemia (Infections and infestations) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 2 | 2
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0
Empyema (Infections and infestations) | 3 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 2
Iliac artery occlusion (Vascular disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lung abscess (Infections and infestations) | 2 | 1
Major depression (Psychiatric disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Pneumocystis test positive (Investigations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 | 20
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 5 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.